CLINICAL TRIAL: NCT03026790
Title: Comparative Effectiveness of Patient-Centered Strategies to Improve Pain Management and Opioid Safety for Veterans
Brief Title: Veterans' Pain Care Organizational Improvement Comparative Effectiveness Study
Acronym: VOICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: OPD-1511-33052
Record Dates: First submitted 2017-01-01; First posted 2017-01-20 (Estimated); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain
Keywords: Opioid analgesics; Opioid partial agonists; Health care delivery; Back pain; Osteoarthritis; Veterans health
MeSH Terms: conditions — Chronic Pain; Back Pain; Osteoarthritis | interventions — Medication Therapy Management; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Telecare collaborative management (TCM) (Active Comparator): Uses medication management approach delivered by a clinical pharmacist care manager with a collaborating physician to address common barriers to effective pain medication management in primary care.
  Interventions: Other: Medication management
- Integrated pain team (IPT) (Active Comparator): Uses a biopsychosocial management approach delivered by a multidisciplinary team that emphasizes non-pharmacological pain management options.
  Interventions: Other: Medication management; Other: Non-pharmacological pain management
- Standard taper options (Active Comparator): The standard taper options arm uses patient education and shared decision-making to guide opioid medication management.
  Interventions: Other: Medication management
- Expanded taper options (Active Comparator): The expanded taper options arm uses patient education and shared decision-making to guide opioid medication management and includes the additional option of rotation to buprenorphine-naloxone.
  Interventions: Other: Medication management; Drug: Buprenorphine-Naloxone

INTERVENTIONS:
Other: Medication management — Individualized management of medications for pain
Other: Non-pharmacological pain management — Individualized management of non-medication pain treatment approaches
  Arms: Integrated pain team (IPT)
Drug: Buprenorphine-Naloxone — Option of using buprenorphine-naloxone to assist with opioid dose reduction or discontinuation
  Arms: Expanded taper options

SUMMARY:
Background and significance: Treatment with opioid pain medications (like hydrocodone and morphine) is common for severe pain, but studies show these medications may not always help and can cause serious problems. High daily doses of opioids can be especially unsafe. To help patients with chronic pain have better quality of life and avoid medication toxicity, health care teams need to manage pain while helping patients reduce opioid medication doses to safer levels.

DETAILED DESCRIPTION:
Study aims: This study will test which of two pain treatment strategies is better for managing pain and helping patients improve safety of opioid medication. For patients on high opioid doses who want to reduce, this study will also test whether offering an extra option for tapering (buprenorphine-naloxone) helps them succeed. Finally, the study will examine patients' and clinicians' experiences with the interventions.

Study description: The study will compare two treatment strategies among patients with pain who are taking long-term opioid pain medications prescribed by VA healthcare facilities across the country. Patients who wish to enter the study will be assigned by chance to telecare collaborative management (TCM) or integrated pain team (IPT). TCM involves a pharmacist and supervising physician working together to find the best medication options for each individual patient. In IPT, a team of clinicians focuses on non-medication pain management options, in addition to pain medication.

All participants will be asked to stay in the study for 12 months. Patients for whom it would be unsafe to participate will not be invited to join. With either treatment strategy, TCM or IPT, participants will have individualized pain care tailored to their needs and preferences. Participants on high opioid medication doses who want to reduce their opioid medication dose will be assigned by chance to get either a regular step-wise taper or a choice between a regular taper or switching to a different medication (buprenorphine-naloxone).

At the end of the study, the two treatment strategies will be compared to see which worked better to (1) decrease pain severity and (2) reduce opioid medication dose. Other outcomes important to patients will also be tracked. These include quality of life, sleep, fatigue, depression, anxiety, and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or high-dose long-term opioid therapy (≥ 20 ME mg daily for at least 3 months) for chronic pain
* Chronic pain of at least moderate severity (defined as pain that is present every or nearly every day for ≥ 6 months and with a score on the PEG 3-item pain measure of ≥ 5)

Exclusion Criteria:

* Dementia diagnosis
* Unstable or severe untreated psychiatric disorder, including severe untreated substance use disorder or active suicidal ideation
* Unstable or end-stage medical disease that would interfere with participation, including cancer requiring active treatment and life expectancy < 12 months
* Documentation of suspected controlled substance diversion
* Inability to communicate by telephone

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing procedures have not been finalized. At a minimum, a complete, cleaned, de-identified copy of the final dataset used in conducting the final analyses of the study will be created and made available within one year after the completion of the study, pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. Depending on feasibility and guidance from VA Office of Research Oversight, a Limited Dataset (LDS) may be created and shared. We have not yet determined how to operationalize data sharing for this study. In the interim, contact the PI for questions or requests.

REFERENCES:
- [Derived] Becker WC, Seal KH, Nelson DB, DeRonne BM, Kats AM, Morasco BJ, Frank JW, Makris UE, Painter JT, Allen KD, Mixon AS, Bohnert A, Reznik TE, Hagedorn HJ, Hammett P, Borsari B, Baxley C, Krebs EE; VOICE Study Group. Buprenorphine, Pain, and Opioid Use in Patients Taking High-Dose Long-Term Opioids: A Randomized Clinical Trial. JAMA Intern Med. 2025 Apr 1;185(4):372-381. doi: 10.1001/jamainternmed.2024.8361. PMID 39960730
- [Derived] Krebs EE, Becker WC, Nelson DB, DeRonne BM, Jensen AC, Kats AM, Morasco BJ, Frank JW, Makris UE, Allen KD, Naylor JC, Mixon AS, Bohnert A, Reznik TE, Painter JT, Hudson TJ, Hagedorn HJ, Manuel JK, Borsari B, Purcell N, Hammett P, Amundson EC, Kerns RD, Barbosa MR, Garvey C, Jones EJ, Noh MY, Okere JB, Bhushan S, Pinsonnault J, Williams BE, Herbst E, Lagisetty P, Librodo S, Mapara PS, Son E, Tat C, Marraffa RA, Seys RL, Baxley C, Seal KH; VOICE Study Group. Care Models to Improve Pain and Reduce Opioids Among Patients Prescribed Long-Term Opioid Therapy: The VOICE Randomized Clinical Trial. JAMA Intern Med. 2025 Feb 1;185(2):208-220. doi: 10.1001/jamainternmed.2024.6683. PMID 39652356
- [Derived] Krebs EE, Becker WC, Nelson D, DeRonne BM, Nugent S, Jensen AC, Amundson EC, Manuel JK, Borsari B, Kats AM, Seal KH. Design, methods, and recruitment outcomes of the Veterans' Pain Care Organizational Improvement Comparative Effectiveness (VOICE) study. Contemp Clin Trials. 2023 Jan;124:107001. doi: 10.1016/j.cct.2022.107001. Epub 2022 Nov 13. PMID 36384218

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: Telecare Collaborative Management (TCM): Uses medication management approach delivered by a clinical pharmacist care manager with a collaborating physician to address common barriers to effective pain medication management in primary care.
- Active Comparator: Integrated Pain Team (IPT): Uses a biopsychosocial management approach delivered by a multidisciplinary team that emphasizes non-pharmacological pain management options.
Period: Overall Study
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Started | 411 | 409
Completed | 358 | 363
Not Completed | 53 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT) | Total
Number analyzed (Participants) | 411 | 409 | 820
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (10.8) | 62.2 (10.4) | 62.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 51 | 111
  Male | 351 | 358 | 709
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 10 | 16
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 63 | 67 | 130
  White | 312 | 297 | 609
  More than one race | 22 | 22 | 44
  Unknown or Not Reported | 4 | 12 | 16

OUTCOME MEASURES:

1. Primary Outcome: Pain Response
Description: Binary response variable defined by reduction of at least 30% in Brief Pain Inventory (BPI) total score from baseline
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 350 | 362
Participants | 58 | 54

2. Secondary Outcome: 50% Reduction in Opioid Daily Dose
Description: Binary response variable defined by reduction of at least 50% in opioid daily dose (morphine-equivalent mg) from baseline
Time Frame: 12 months
Population: All participants who were alive at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 403 | 399
Participants | 102 | 98

3. Secondary Outcome: Composite Response
Description: Binary composite response variable defined by achieving at least a 30% reduction in BPI total score and at least 50% reduction in opioid daily dose from baseline.
Time Frame: 12 months
Population: All participants who completed the measure at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 350 | 362
Participants | 17 | 17

4. Secondary Outcome: Brief Pain Inventory (BPI) Total Score
Description: Brief Pain Inventory (BPI) total score calculated as average of 11 items (range 0-10; higher is worse)
Time Frame: 12 months
Population: All participants who completed the measure at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 351 | 362
units on a scale | 6.07 (1.81) | 6.01 (1.91)

5. Other Pre Specified Outcome: VR-12 Physical Component Score
Description: Veterans RAND 12-item health survey (VR-12) Physical Component Score (range 0-100; higher is better)
Time Frame: 12 months
Population: All participants who completed the measure at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 357 | 363
units on a scale | 41.9 (12.9) | 42.5 (13.2)

6. Other Pre Specified Outcome: Symptom Checklist
Description: Medication-related adverse symptoms count (0-19; higher is worse)
Time Frame: 12 months
Population: All participants who completed the measure at 12 months
Measure: Mean (Standard Deviation); unit: symptom count
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 270 | 278
symptom count | 4 (3.7) | 3.5 (3.5)

7. Other Pre Specified Outcome: PODS Problems
Description: Prescribed Opioids Difficulty Scale (PODS) Problems score (range 0-32; higher is worse)
Time Frame: 12 months
Population: All participants who completed the measure at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 234 | 245
units on a scale | 3.4 (6.2) | 2.5 (5.1)

8. Other Pre Specified Outcome: PHQ-8
Description: Patient Health Questionnaire 8-item (PHQ-8) depression scale score (range 0-24; higher is worse)
Time Frame: 12 months
Population: All participants who completed the measure at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 320 | 327
units on a scale | 8.79 (5.84) | 5.2 (5.85)

9. Other Pre Specified Outcome: GAD-7
Description: General Anxiety Disorders 7-item questionnaire (GAD-7) score (range 0-21; higher is worse)
Time Frame: 12 months
Population: All participants who completed the measure at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 319 | 326
units on a scale | 6.01 (5.61) | 5.55 (5.61)

10. Other Pre Specified Outcome: PROMIS Sleep Disturbance
Description: Patient Reported Outcomes Measurement Information System (PROMIS) sleep disturbance short-form 4a T-score (higher is worse). Raw scores were rescaled into standardized T-scores with a mean of 50 representing the average for the US population and a standard deviation (SD) of 10. A person with a T-score of 40 is one SD below the mean.
Time Frame: 12 months
Population: All participants who completed the measure at 12 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 310 | 322
T-score | 57.2 (9.1) | 55.5 (9.3)

11. Other Pre Specified Outcome: PROMIS Fatigue
Description: Patient Reported Outcomes Measurement Information System (PROMIS) fatigue short-form 4a T-score (higher is worse). Raw scores were rescaled into standardized T-scores with a mean of 50 representing the average for the US population and a standard deviation (SD) of 10. A person with a T-score of 40 is one SD below the mean.
Time Frame: 12 months
Population: All participants who completed the measure at 12 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 310 | 321
T-score | 57.1 (10.9) | 55.7 (11.1)

12. Other Pre Specified Outcome: Headache Impact Test
Description: Headache Impact Test score (range 36-78; higher is worse)
Time Frame: 12 months
Population: All participants who completed the measure at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 289 | 303
units on a scale | 50.77 (12.26) | 49.84 (11.54)

13. Other Pre Specified Outcome: VR-12 Mental Component Score
Description: Veterans RAND 12-item health survey (VR-12) Mental Component Score (range 0-100; higher is better)
Time Frame: 12 months
Population: All participants who completed the measure at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 356 | 363
units on a scale | 41.9 (12.9) | 42.5 (13.2)

14. Other Pre Specified Outcome: PODS Concerns
Description: Prescribed Opioids Difficulty Scale (PODS) Concerns score (range 0-28; higher is worse)
Time Frame: 12 months
Population: All participants who completed the measure at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
Number analyzed (Participants) | 244 | 254
units on a scale | 3.8 (4.7) | 4 (4.8)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Active Comparator: Telecare Collaborative Management (TCM) | Active Comparator: Integrated Pain Team (IPT)
All-Cause Mortality (participants affected / at risk) | 7/358 | 9/363
Serious Adverse Events (participants affected / at risk) | 109/358 | 109/363
Other Adverse Events (participants affected / at risk) | 207/358 | 178/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator: Telecare Collaborative Management (TCM) (N=358) | Active Comparator: Integrated Pain Team (IPT) (N=363)
Hospitalization (General disorders) | 109 | 109
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator: Telecare Collaborative Management (TCM) (N=358) | Active Comparator: Integrated Pain Team (IPT) (N=363)
Emergency department visit (General disorders) | 207 | 178

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03026790/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT03026790/ICF_001.pdf